CLINICAL TRIAL: NCT05720715
Title: Evaluation of the Safety and Efficacy of Cyclosporine A 0.05% Eye Drops in Management of Non- Necrotizing Herpetic Stromal Keratitis; a Prospective Controlled Clinical Trial
Brief Title: Clinical Outcomes of Cyclosporine Eye Drops in Management of Herpetic Keratitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Farwaniya Hospital (Other Government)
Responsible Party: Principal Investigator, Nancy Lotfy, MD, Dr, Farwaniya Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7080
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Outcomes of Cyclosporine Eye Drops in Herpetic Keratitis
MeSH Terms: interventions — Cyclosporine; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): receive cyclosporine eye drops together with prednisolone eye drops.
  Interventions: Drug: cyclosporine A 0.05% eye drops
- group B (Placebo Comparator): receive topical prednisolone with placebo eye drops (tear replacement).
  Interventions: Drug: cyclosporine A 0.05% eye drops

INTERVENTIONS:
Drug: cyclosporine A 0.05% eye drops — Patients diagnosed with herpetic stromal keratitis are randomly divided into 2 groups; Group A: receive cyclosporine eye drops together with prednisolone eye drops.
  Group B: receive topical prednisolone with placebo eye drops (tear replacement).
  The 2 groups receive systemic acyclovir therapeutic dose 400 mg five times daily, which then tapered to twice daily prophylactic dose after one month of treatment. Follow up for patients is scheduled as a weekly visit for a duration of 2 months.

SUMMARY:
Objective: To compare the additive effect of topical cyclosporine A 0.05% eye drops to prednisolone eye drops, with topical prednisolone acetate 1% eye drops alone in treatment of herpetic stromal keratitis.

Methods: Patients diagnosed with herpetic stromal keratitis are randomly divided into 2 groups; Group A: receive cyclosporine eye drops together with prednisolone eye drops.

Group B: receive topical prednisolone with placebo eye drops (tear replacement).

The 2 groups receive systemic acyclovir therapeutic dose 400 mg five times daily, which then tapered to twice daily prophylactic dose after one month of treatment. Follow up for patients is scheduled as a weekly visit for a duration of 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with herpetic stromal keratitis

Exclusion Criteria:

* associated ocular diseases, DM, renal disease, pregnancy, breast feeding.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
duration of ttt | 3 months
  duration of treatment until complete resolving of keratitis

SECONDARY OUTCOMES:
improvement in visual acuity | 3 months
  by snellen chart

CONTACTS AND LOCATIONS:
Overall Officials: Salah Al-rasheedy, MD, Study Chair — Farwaniya Hospital
Locations (1):
- Farwanyia Hospital, Al Farwānīyah, Farwanyia, Kuwait